CLINICAL TRIAL: NCT07047391
Title: Prediction of Pulmonary Problems in Individuals With Rheumatoid Arthritis-Associated Interstitial Lung Disease
Brief Title: Prediction of Pulmonary Problems
Status: Completed | Type: Observational
Sponsor: Zülal TATAR (Other)
Responsible Party: Sponsor-Investigator, Zülal TATAR, Researcher, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: Pulmonary Problem
Record Dates: First submitted 2025-06-20; First posted 2025-07-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Muscle Strength; Oxygen Saturation; Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to examine the relationship between respiratory muscle strength and grip strength, muscle strength, oxygen saturation of peripheral muscles, dyspnea and respiration, cough, and health-related quality of life in individuals with Interstitial Lung Disease Associated with Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* ≥18 individuals diagnosed with RA by the same rheumatologist based on published results

Exclusion Criteria:

* Individuals with >10 pack-year smoking history
* Severe functional limitations
* Cardiopulmonary and/or neurological disease unrelated to RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis-associated interstitial lung disease follow-up at Pamukkale University Hospital
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of respiratory muscle strength | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  One of the most commonly used and noninvasive methods for assessing respiratory muscle strength is the measurement of MIP and MEP. Respiratory muscle strength was measured using a portable, electronic, oral pressure measuring device (Micro Medical MicroMPM, UK). These are intraoral pressures measured during maximal inspiration against a valve that closes the airway during maximum inspiration and expiration.
Oxygen Saturation Measurement | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  Oxygen saturation measurement was performed with the MOXY (Fortiori Design LLC., Minnesota, USA) device. MOXY is a medical device with dimensions of 61x44x21 mm and a weight of 42 gr. It is an infrared measurement device called "near infrared spectroscopy" that measures oxygen saturation and total hemoglobin in muscle capillaries.

SECONDARY OUTCOMES:
Modified Borg Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  Although it is frequently used today to define the severity of exertional dyspnea, it is a scale that can also be used to evaluate the severity of resting dyspnea. It consists of ten items that define the severity of dyspnea according to their degrees. Scoring is done between 0 (not at all) and 10 (very severe).
Modified Medical Research Council Dyspnea Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  It is a scale based on various physical activities that cause dyspnea. It consists of five items. The patient rates respiratory distress between 0 (no shortness of breath) and 4 (shortness of breath during activities such as being homebound and dressing).
Visual Analog Scale | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  It consists of a 100 mm long horizontal line with the words "none" and "very severe" written on one end. The patient marks the severity of the current respiratory distress on the line using these two degrees as criteria. Scoring is done by measuring the marked area with the help of a tape measure.
Leicester Cough Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  Measures the effect of cough on quality of life. It consists of 19 questions. It has psychological, social and physical sub-dimensions. The cut-off value of the scale is not defined; low scores indicate greater effect from cough, i.e. worse quality of life. The total severity score ranges from 3 to 21.
St. George's Respiratory Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  It will be used to evaluate the health-related quality of life of the cases. SGRQ consists of three categories where the symptoms, activities and the effects of the disease on their daily lives are evaluated. The symptoms examined are cough, sputum, wheezing and shortness of breath. Physical functions, housework and hobbies are questioned to determine the activity status. These are activities limited by shortness of breath. The survey consisting of a total of 76 questions is completed in 20 minutes. There is an evaluation scale between zero and 100 points. Zero indicates perfect health status, 100 indicates the worst health status.
Short Form-36 Quality of Life Survey | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  Short form-36 is a quality of life scale consisting of 36 items that can be filled by the patient and whose validity and reliability have been shown in studies in patients with musculoskeletal disorders. The Turkish version of SF-36 was used in our study. This scale includes 8 separate health-related headings as physical function (10 items), social function (2 items), physical role limitation (4 items), emotional role limitation (3 items), mental health (5 items), vitality (4 items), pain (2 items), general health (6 items).
Health Assessment Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  Since it evaluates activities of daily living comprehensively and in all dimensions, HAQ was preferred in our study to assess the disability level. It includes 20 questions across 8 domains (dressing, arising, eating, walking, hygiene, reach, grip, and common activities). Each question is scored between 0 and 3 (without any difficulty = 0, with some difficulty = 1, with much difficulty = 2, unable to do = 3). The highest score of each subsection is summed up and divided by 8 to determine the total score between 0 and 3. A high score indicates a low functional level
Disease Activity | Evaluations started immediately after receiving ethics committee approval and will be completed within 1 months, which is the study period.
  Disease activity in rheumatoid arthritis will be assessed using the Clinical Disease Activity Index (CDAI). This index is calculated based on four main parameters: the number of painful joints, the number of swollen joints, the visual analog scale of global disease activity as assessed by the patient, and the visual analog scale of global disease activity as assessed by the physician. CDAI scores of 0-2.8 indicate remission, 2.9-10 indicate low disease activity, 11-22 indicate moderate activity, and 22-76 indicate high activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)